CLINICAL TRIAL: NCT05731648
Title: Role of Functional Neurosurgery in Management of Spasticity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Zanaty, Assistant lecturer, Assiut University
Other Study IDs: Neurosurgery and spasticity
Record Dates: First submitted 2023-01-30; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Functional Neurological Disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intrathecal balofen pump — Management of spasticity
  Other Names: spinal cord stimulator

SUMMARY:
Spasticity can result from a variety of causes in neural axis from which most common are cerebral palsy, strokes, cerebral haemorrhage, multiple sclerosis , traumatic brain injury and spinal cord injury and underlying mechanism is broadly due to decrease inhibition of the spinal network.

Clinical evaluation for spasticity involve series of clinical assessment , physical examination , and neurophysiological testing. quantitative evaluation of spasticity can be measured using modified Ashworth scale which is the most widely used clinical spasticity scale and can be used for various clinical conditions causing spasticity

DETAILED DESCRIPTION:
Currently, the management of spasticity spans in a continuum between non-invasive and invasive intervention to modulate its effects and improve patients' Quality of life and when spasticity becomes excessive and aggravates disability, functional neurosurgery can be a resource.

Neurosurgical procedures for management of spasticity are classified according to whether their effect is generalized or focal and whether they are reversible or irreversible. Procedures include intrathecal baclofen pump , spinal cord stimulation and lesioning techniques peripheral nerves , dorsal roots , spinal cord or dorsal root entry zone

ELIGIBILITY:
Inclusion Criteria:

* Patients with spasticity refractory to medical treatment (most commonly administered oral medications for managing spasticity are diazepam, dantrolene sodium, and baclofen) and physiotherapy

Exclusion Criteria:

* Patients unfit for neurosurgical intervention

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Spasticity
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and efficacy of neurosurgical procedures | 6 month
  Rate of complication ( infection , bleeding , Device Malware )
Evaluate Changes in Modified Ashworth scale | 6 month
  * 0: No increase in muscle tone
  * 1: Slight increase in muscle tone, with a catch and release or minimal resistance at the end of the range of motion when an affected part(s) is moved in flexion or extension
  * 1+: Slight increase in muscle tone, manifested as a catch, followed by minimal resistance through the remainder (less than half) of the range of motion
  * 2: A marked increase in muscle tone throughout most of the range of motion, but affected part(s) are still easily moved
  * 3: Considerable increase in muscle tone, passive movement difficult
  * 4: Affected part(s) rigid in flexion or extension

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hinderer SR, Dixon K. Physiologic and clinical monitoring of spastic hypertonia. Phys Med Rehabil Clin N Am. 2001 Nov;12(4):733-46. PMID 11723863
- [Result] Kheder A, Nair KP. Spasticity: pathophysiology, evaluation and management. Pract Neurol. 2012 Oct;12(5):289-98. doi: 10.1136/practneurol-2011-000155. PMID 22976059